CLINICAL TRIAL: NCT06260748
Title: A Phase 3, Prospective, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Chenodeoxycholic Acid (CDCA), With an Open-Label Cohort, in Newly Diagnosed Participants With Cerebrotendinous Xanthomatosis (CTX)
Brief Title: A Study of Chenodeoxycholic Acid (CDCA) in Newly Diagnosed Participants With Cerebrotendinous Xanthomatosis (CTX)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBI-CDCA-001; 2023-505759-29-00 (Other: EU Clinical Trials Register)
Record Dates: First submitted 2024-02-01; First posted 2024-02-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cerebrotendinous Xanthomatoses
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 Diarrhea-Evaluable (Experimental): Diarrhea-evaluable participants aged 12-75 years old who did not use continence aids that precluded assessment or evaluation of stool frequency and consistency during the screening/baseline period; randomized 1:1 to receive either placebo or CDCA.
  Interventions: Drug: Chenodeoxycholic acid; Drug: Chenodeoxycholic acid Placebo
- Group 2a Non-Diarrhea Evaluable (Active Comparator): Non-diarrhea-evaluable participants aged 12-75 years old who do not have stable, clinically burdensome diarrhea or their diarrhea cannot be fully characterized.
  Interventions: Drug: Chenodeoxycholic acid
- Group 2b Pediatrics (Active Comparator): Participants aged 2 to less than 12 years old with or without clinically burdensome diarrhea.
  Interventions: Drug: Chenodeoxycholic acid

INTERVENTIONS:
Drug: Chenodeoxycholic acid — 250mg capsules
  Other Names: CDCA
Drug: Chenodeoxycholic acid Placebo — Placebo to match
  Arms: Group 1 Diarrhea-Evaluable

SUMMARY:
This study is designed to demonstrate the beneficial effect of CDCA in the treatment of CTX-associated diarrhea in approximately 10 participants aged 2-75 years old with newly diagnosed CTX or suspected CTX who have never received treatment with CDCA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (or assent form as appliable)
* Aged from 2 to 75 years old
* Has a new or suspected diagnosis of CTX as defined by an elevated plasma cholestanol concentration (>10 mg/L/>25.7 μmol/L) in conjunction with a clinical presentation consistent with the diseased as assessed by the investigator
* Has never received treatment with CDCA
* Has never received treatment with other bile acid products

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator, precludes the participant's participation in the study
* Presence of known hepatocyte dysfunction or bile ductal abnormalities such as intrahepatic cholestasis, primary biliary cirrhosis or sclerosing cholangitis
* Inability to adhere to treatment and visit schedule
* Female participants who are pregnant
* Female participants who are breast feeding
* Female participants who are using estrogen-containing compounds and cannot/will not discontinue them for the duration of the study
* Female participants of childbearing potential who are not using locally approved birth control method(s) or double barrier contraception (ie, condom and diaphragm, condom or diaphragm and spermicidal gel or foam)
* Taking any of the following medications: bile acid products; inhibitors of bile acid transporters; bile acid binding resins; aluminum-based antacids; coumarin and its derivatives; cholestyramine; ciclosporin; sirolimus; or phenobarbital

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at Week 4 in average number of stools with a BSS score of 6 or 7 per day | Up to 4 weeks

SECONDARY OUTCOMES:
Change in plasma cholestanol levels from baseline to Week 12 | Up to 12 weeks
  All groups combined
Change in urine and/or plasma bile alcohol levels from baseline to Week 12 | Up to 12 weeks
  All groups combined
Incidence of, severity/intensity of, and relationship to study drug of AEs | Up to 20 weeks
Incidence of, severity/intensity of, and relationship to study drug of SAEs | Up to 20 weeks
Incidence of, severity/intensity of AESIs | Up to 20 weeks
  Diarrhea and hepatic dysfunction
Incidence of, severity/intensity of, and changes in laboratory values | Up to 20 weeks
Incidence of, severity/intensity of, and changes in physical examination | Up to 20 weeks
Incidence of, severity/intensity of, and changes in vital signs | Up to 20 weeks
Number of participants with discontinuations due to AEs | Up to 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel